CLINICAL TRIAL: NCT01214278
Title: Relative Bioavailability of Different n-3 Fatty Acid Formulations in Humans
Brief Title: Bioavailability of Different n-3 Fatty Acid Formulations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gottfried Wilhelm Leibniz Universität Hannover (Other)
Responsible Party: Principal Investigator, M. Sc. Simone Schmidt, Master of Science, Gottfried Wilhelm Leibniz Universität Hannover
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GWLUH-002; GWLUH2010 (Other: 02)
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Health
Keywords: bioavailability; marine n-3 fatty acids; EPA; DHA
MeSH Terms: interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Supplement 1 (Experimental): EPA+DHA as re-esterified triglycerides (rTGs) from fish-oil uncoated capsules
  Interventions: Drug: rTG
- Supplement 2 (Experimental): EPA+DHA as rTGs from fish-oil in gastric acid resistant (coated) capsules (GArTG)
  Interventions: Drug: GArTG
- Supplement 3 (Experimental): EPA+DHA as ethylesters (EE) from fish-oil uncoated capsules
  Interventions: Drug: EE
- Supplement 4 (Experimental): DHA+EPA as phospholipids from krill-oil, uncoated capsules (KPL)
  Interventions: Drug: KPL

INTERVENTIONS:
Drug: rTG — EPA+DHA as re-esterified triglycerides (rTGs) from fish-oil; uncoated capsules (4 per day); 2016 mg n3 fatty acids daily (1008 mg EPA and 672 mg DHA)
  Other Names: re-esterified triglycerides
  Arms: Supplement 1
Drug: GArTG — EPA+DHA as rTGs from fish-oil in gastric acid resistant (coated) capsules (GArTG); 4 capsules per day; 2016 mg n-3 fatty acids (1008 mg EPA and 672 mg DHA)
  Other Names: rTG in gastric acid resistant capsules
  Arms: Supplement 2
Drug: EE — EPA+DHA as ethylesters (EE) from fish-oil uncoated capsules (4 per day); 2016 mg n-3 fatty acids (1008 mg EPA and 672 mg DHA)
  Other Names: ethylesters
  Arms: Supplement 3
Drug: KPL — DHA+EPA as phospholipids from krill-oil, uncoated capsules (KPL); 7 capsules per day; 2100 mg n-3 fatty acids (1050 mg EPA and 630 mg DHA)
  Other Names: phospholipids from krill-oil
  Arms: Supplement 4

SUMMARY:
The aim of this study is to examine differences in short term bioavailability between four n-3 FA formulations in healthy males.

DETAILED DESCRIPTION:
The long-chain n-3 fatty acids (n-3 FAs) eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are known to positively affect the lipid profile, vascular tone and blood coagulation. Moreover, EPA and DHA possess anti-inflammatory effects and play a central role in the functioning of the brain and central nervous system. Therefore, an increased EPA and DHA intake is highly recommend. However, it is unknown whether different chemical formulations of EPA + DHA rich supplements (re-esterified triglycerides, ethyl-esters, phospholipids) have identical bioavailability. The objective of this study is to examine differences in short term bioavailability between four n-3 FA formulations:

* Supplement 1: EPA+DHA as re-esterified triglycerides (rTGs) from fish-oil uncoated capsules
* Supplement 2: EPA+DHA as rTGs from fish-oil in gastric acid resistant (coated) capsules (GArTG)
* Supplement 3: EPA+DHA as ethylesters (EE) from fish-oil uncoated capsules
* Supplement 4: DHA+EPA as phospholipids from krill-oil, uncoated capsules (KPL)

The study preparations are certificated supplements and available on the market.

There are no comparative investigations, which analyzed the bioavailability of these four n-3 FA formulations in a similar design.

ELIGIBILITY:
Inclusion Criteria:

* males,
* 20-50 years,
* Caucasian,
* healthy,
* body mass index (BMI) 20-28 kg/m²,
* no medical treatment,
* written confirmation of the subjects after detailed spoken and written explanation about the study contents,
* ability and willingness of the participants to attend the investigator's orders (compliance of the study conditions, consumption of the study drugs according to the dosage commendation

Exclusion Criteria:

* medical treatment (especially corticosteroids, anti-inflammatory drugs, blood lipids lowering drugs (e.g. statines, fibrates, bile acid exchanger resin, phytosterols)
* taking any supplements with n-3 FAs, phytosterols, polyglucosamines (Chitosan) or other lipid binding ingredients
* daily consumption of n-3 FAs rich fish (salmon, mackerel, herring)
* heavy chronic diseases (tumors, diabetes typ 1, etc.), documented heart disease, documented blood clotting disorders, renal failure, liver diseases
* documented blood clotting disorders and consumption of coagulation-inhibiting drugs (for example Marcumar, ASS)
* allergy or intolerance to fish/fish oil or any of the study ingredients of the test products
* chronic gastro-intestinal diseases (Colitis ulcerosa, Morbus Crohn, pancreatic insufficiency)
* donation of blood in the last 6 weeks
* routine consumption of laxative
* alcohol-, drug- and/or medicament dependence
* subjects who are not in agreement with the study conditions
* refusal or rather reset of the consent from the subject
* active participation in other investigational drug or device trial within the last 30 days

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under concentration time curve (AUC) | about 24 hours
  Concentration of eicosapentanoiec acid (EPA) and docosahexanoiec acid (DHA) was measured at baseline and after 2, 4, 6, 8 and 24 hours.

SECONDARY OUTCOMES:
Area under concentration time curve (AUC) | about 48 and 72 hours
  Concentration of eicosapentanoiec acid (EPA) and docosahexanoiec acid (DHA) was measured at baseline and after 2, 4, 6, 8, 24, 48 and 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hahn, Prof., Study Director — Gottfried Wilhelm Leibniz University of Hanover
Locations (1):
- Gottfried Wilhelm leibniz University of Hanover, Hanover, Lower Saxony, Germany

REFERENCES:
- See also: web page of the institute — http://www.nutrition.uni-hannover.de